CLINICAL TRIAL: NCT06184568
Title: A Multicenter, Randomized, Open-label Phase 3 Study Comparing the Efficacy and Safety of IBI362 Versus Semaglutide in Chinese Participants With Early Type 2 Diabetes and Obesity (DREAMS-3)
Brief Title: A Study Comparing IBI362 vs Semaglutide in Chinese Adults With Early Type 2 Diabetes and Obesity
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIBI362A303
Record Dates: First submitted 2023-12-14; First posted 2023-12-28 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — mazdutide; semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semaglutide (Active Comparator)
  Interventions: Drug: Semaglutide
- IBI362 (Experimental)
  Interventions: Drug: IBI362

INTERVENTIONS:
Drug: IBI362 — Once-weekly injections of gradually increased doses of IBI362, subcutaneously (SC)，starting dose is IBI362 2.0 mg, continuous After 4 weeks of administration, increase to IBI362 4.0 mg. After 4 weeks of continuous administration, continue to increase to IBI362.
  Arms: IBI362
Drug: Semaglutide — Once-weekly injections of gradually increased doses of Semaglutide, subcutaneously (SC)，starting dose is semaglutide 0.25mg, after 4 weeks of continuous administration, increase to semaglutide 0.5mg, after 4 weeks of continuous administration, continue Upgrade to semaglutide 1.0 mg for 24 weeks.
  Arms: Semaglutide

SUMMARY:
This is a multicenter, randomized, Open-label Phase 3 clinical study comparing the efficacy and safety of IBI362 6 mg OW versus Semalgutide 1 mg OW in obese(BMI≥28kg/m2) early T2D subjects. Subjects will be randomly assigned to IBI362 6 mg and Semalgutide 1 mg groups for 32 weeks (active-controlled treatment period). In the extension period, participants originally on mazdutide were assigned to continue for an additional 24 weeks with mazdutide 9 mg or 6 mg based on whether they achieved the weight-loss target. All study treatment will be administered once-weekly and subcutaneously. The entire trial cycle includes a 2-week screening period, a 32-week active-controlled treatment period, a 24 week extension period and a 4-week drug withdrawal safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 years or older at the time of signing informed consent
* T2D was diagnosed according to WHO standards in 1999(≤5 years)
* The blood glucose was not well controlled after diet and exercise with/without sable metformin(≥1500mg/day，no more than 2550mg/day) within 3 months before screening, and the local laboratory tested 7.5% ≤ HbA1c ≤9.5% during screening
* Have a BMI ≥28 kg/m2

Exclusion Criteria:

* Subjects who the investigator thinks may be allergic to the components in the study drug or similar drugs
* A self-reported change in body weight above 5% within 3 months before screening
* Oral hypoglycemic drugs other metformin have been used within 2 months before screening.
* Previous diagnosis of type 1 diabetes (including adult latent autoimmune diabetes)
* There are active or untreated malignant tumors within 5 years before screening, or patients are in remission of clinical malignant tumors (except patients with skin basal cell carcinoma and squamous cell carcinoma, cervical carcinoma in situ, prostate carcinoma in situ or papillary thyroid carcinoma who have no recurrence after surgery)
* Mental illness existed in the past or at the time of screening, and the researcher thinks it is not suitable to participate in this study
* Pregnant or lactating women, or men or women who are fertile and unwilling to use contraception throughout the study period
* The investigator believes that the subject has any other factors that may affect the efficacy or safety evaluation of this study and is not suitable to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2024-02-29 (Actual); Primary Completion 2026-02-09 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects who achieve composite endpoint of HbA1c <7.0% and ≥10% weight loss | Week 32

SECONDARY OUTCOMES:
Proportion of subjects who achieve composite endpoint of HbA1c <7.0% and ≥15% weight loss | Week 32
Proportion of subjects who achieve composite endpoint of HbA1c <7.0% and ≥5% weight loss | Week 32
Proportion of subjects who achieve composite endpoint of HbA1c<6.5% and ≥5%, ≥10% or ≥15% weight loss | Week 32
Change from Baseline in HbA1c | Week 32
Change from Baseline in Fasting Plasma Glucose | Week 32
Proportion of subjects who achieve composite endpoint of HbA1c <7.0%，≤6.5% or <5.7% | Week 32
Percent Change from Baseline in Body Weight | Week 32
Change from Baseline in Waist Circumference | Week 32
Proportion of subjects who achieve ≥5%, ≥10% or ≥15% weight loss | Week 32
Change from Baseline in Blood Pressure(Systolic and Diastolic) | Week 32
Percent Change from Baseline in Triglycerides, Total Cholesterol, LDL-c, HDL-c, non-HDL-c | Week 32

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China